CLINICAL TRIAL: NCT01204255
Title: Absorption of "ABH Gel" (Ativan®, Lorazepam; Benadryl®, Diphenhydramine; and Haldol®, Haloperidol Gel) From the Skin of Normal Volunteers
Brief Title: Lorazepam, Diphenhydramine Hydrochloride, and Haloperidol Gel in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-13108; NCI-2010-01968 (Registry Identifier: CTRP); PEP-10-174-1-PCSM (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: healthy, no evidence of disease
MeSH Terms: interventions — Lorazepam; Diphenhydramine; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients apply lorazepam, diphenhydramine hydrochloride, and haloperidol gel topically over 2 minutes.
  Interventions: Drug: lorazepam; Drug: diphenhydramine hydrochloride; Drug: haloperidol; Other: questionnaire administration; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lorazepam — Given topically
  Other Names: Ativan
Drug: diphenhydramine hydrochloride — Given topically
  Other Names: Benadryl; Bendylate; Eldadryl; SK-Diphenhydramine
Drug: haloperidol — Given topically
  Other Names: Haldol; McN-JR-1625; R-1625
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Lorazepam, diphenhydramine hydrochloride, and haloperidol gel, when absorbed into the skin, may be an effective treatment for nausea and vomiting.PURPOSE: This clinical trial studies lorazepam, diphenhydramine hydrochloride, and haloperidol gel in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:I. To study the absorption of the three components in the topical ABH gel in 10 healthy volunteers, and determine if there are any adverse effects. OUTLINE: Patients apply lorazepam, diphenhydramine hydrochloride, and haloperidol gel topically over 2 minutes. After completion of study treatment, patients are followed up for 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Completed a medical screening questionnaire
* English speaking
* No allergies to the drugs
* Able to complete the forms
* If a woman of childbearing age, agree to use contraception

Exclusion Criteria:

* History of substance abuse, psychiatric disorder, acquired brain injury, the possibility of pregnancy (not using birth control, and of child bearing age)
* Use of any medication that would contraindicate benzodiazepine administration
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Smith, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Lorazepam, Diphenyhydramine, Haloperidol Absorption
Description: Level of lorazepam absorption measured by the serum concentration of the drug
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Application of Lorazepam, Diphenhydramine, Haloperidol: Topical application of lorazepam, diphenhydramine, haloperidol
Arm/Group | Application of Lorazepam, Diphenhydramine, Haloperidol
Number analyzed (Participants) | 10
ng/ml
  lorazepam absorption | 0 (0)
  diphenhydramine absorption | .08 (.12)
  haloperidol absorption | 0 (0)

2. Secondary Outcome: Side Effects
Time Frame: 3 months
Measure: Number; unit: Total number of side effects
Arm/Group | Application of Lorazepam, Diphenhydramine, Haloperidol
Number analyzed (Participants) | 10
Total number of side effects | 0

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No